CLINICAL TRIAL: NCT06732700
Title: The Effect of Integrated Neuromuscular Inhibition Technique on Cervical Proprioception in Patients With Forward Head Posture
Brief Title: Effect of INIT on Cervical Proprioception in Patients With Forward Head Posture
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC/01940 Iqra Rashid
Record Dates: First submitted 2024-10-28; First posted 2024-12-13 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Forward Head Posture
Keywords: INIT, Forward Head Posture, Joint Position Error Test

STUDY DESIGN:
Intervention Model Description: Experimental Group: Group A INIT+ Posture Corrective Exercises Control Group: Group B Posture corrective exercise
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group: 1 (Experimental): INIT+ Posture Corrective Exercises INIT consists of Ischemic Compression, Strain-Counter Strain and Muscle Energy Technique. INIT will be performed on Upper Trapezius, Levator Scapulae and Sternocleidomastoid. The patient will be lying supine; First We will identify the TrPs in the muscle. After that the patient will be placed in comfortable position, first technique applied will be Ischemic Compression. The technique will be applied for 90 secs. After this SCS will be applied, moderate digital pressure will maintained over the active TrP as the position of ease will be identified, it will be held for 20-30 s and repeated for three to five repetitions. Lastly, the subjects will receive MET directed towards the involved muscle. Each isometric contraction will be held for 7-10 sec and stretch will be held for 30 seconds and will be repeated three to five times per treatment session.
  Posture corrective exercises given to control group will also be performed
  Interventions: Other: Integrated Neuromuscular Inhibition Technique and Posture Corrective Exercises.
- Control Group: 2 (Active Comparator): Posture corrective exercise Strengthening exercises: a) chin tuck in supine lying with the head in contact with the floor, (1 sets, 10 reps) b) Y-to-I exercise in a prone position (1 sets, 10 reps) c) Prone horizontal abduction with external rotation (1 sets, 10 reps).
  Stretching Exercises:
  d) one-sided unilateral self-stretch of pectoralis minor in standing position (stretch 30 sec, 5 reps) e) static sternocleidomastoid stretch (stretch 30 sec, 5 reps) f) static levator scapulae stretch (stretch 30 sec, 5 reps).
  Interventions: Other: Integrated Neuromuscular Inhibition Technique and Posture Corrective Exercises.

INTERVENTIONS:
Other: Integrated Neuromuscular Inhibition Technique and Posture Corrective Exercises. — INIT will be performed for experimental group and then posture corrective exercises will be performed and for control group only posture corrective exercises will be performed

SUMMARY:
The purpose of the study is to determine the effects of Integrated Neuromuscular Inhibition Technique on Cervical Proprioception in Patients with Forward Head Posture. A randomized control trial was conducted at Riphah International University, Gulberg Green Campus, Islamabad. The sample size was 42 calculated through G-Power. The participants were divided into two interventional groups each having 21 participants. The study duration was six months. Sampling technique applied was Non-probability Purposive sampling for recruitment. Only 18 to 40 years participants with CVA angle less than 50 degree were included in the study. Tools used in this study are Inclinometer, Mobile phone, Labtop, Kinovea Software, NPRS Scale, Laser Beam. Data was collected at Baseline, after 1st session at the end of 2nd week and 4th week. Data analyzed through SPSS version 23.

DETAILED DESCRIPTION:
Forward Head Posture is defined as ≥5 cm in horizontal distance between the tragus of the ear and the posterior angle of acromion in a standing position. The forward head position is characterized by extension of the upper cervical spine (Cl-C3), and flexion of the lower cervical spine (C4-C7), while the cervical curvature is increased. According to study conducted in 2019, Craniovertebral angle is Formed between C7 spinous process and tragus of ear. Forward head posture is present in all age groups, 22-24 years is the mean age group in males with normal CVA about 48.8 degrees, while in females the CVA angle is 47.6 and their mean age is 23-66 years. Normal craniovertebral angle is 49.9 degrees.

Joint position sense is a part of proprioception, which affects body posture and stability. It is influenced by muscle spindles, which respond to changes in muscle length and speed. Forward Head Posture (FHP) causes changes in the lengths of neck muscles, leading to poor joint position sense.

The integrated neuromuscular inhibition technique is one of the manual therapies that are directed to trigger point treatment; this technique consists of ischemic compression, Strain Counter-Strain, and Muscle Energy Technique. Intermittent ischemic pressure increases blood flow, Strain Counter-Strain decreases muscle tone, and Muscle Energy Technique encourages muscle easing, this leads to improvements in pain, function, and range of motion.

A Study in 2019 reported the shortness of Levator scapulae associated with Forward Head Posture leads.

In 2020 Khan et al. carried out research which showed tightness of Sternocleidomastoid muscle in patients with Forward Head Posture.

A study conducted in 2023 evaluated the effect of dry needling of Upper trapezius muscle in Forward Head Posture and results showed one session of dry needle therapy with stretching exercises could improve Pain and Pressure Threshold, Range of Motion, craniovertebral angle, which improved Forward Head Posture.

According to a study conducted in 2020 The craniovertebral angle had a negative correlation with position sensing and individuals with Forward Head Posture had a higher error value when observing cervical position sensing than individual with normal head posture.

According to a study of 2018, integrated neuromuscular inhibition technique is effective in improving cervical function by reducing the trigger points on upper trapezius muscle in mechanical neck pain.

Mustafa et al. in 2023 found that integrated neuromuscular inhibition technique to a multimodal treatment program (Mulligan (SNAG, NAGS) with isometric exercises) improve neck function.

ELIGIBILITY:
Inclusion Criteria:

* Both Male and Female patients
* CVA less than 50 degree
* Age 18-40 years
* Neck pain for more than 3 months
* NPRS > 3
* Decreased Cervical ROMs
* Active trigger points in following muscles (Upper Trapezius, Sternocleidomastoid, Levator Scapulae)

Exclusion Criteria:

* History of cervical or facial trauma or surgery.
* Congenital anomalies of spine such as scoliosis.
* Systemic arthritis.
* Any disorder of Central Nervous System.
* Patients with cognitive deficit

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Estimated)
Dates: Start 2024-04-18 (Actual); Primary Completion 2024-12-22 (Estimated); Study Completion 2024-12-22 (Estimated)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale | 40 minutes session, thrice a week for 4 weeks.
  The NPRS is a segmented numeric version of the visual analog scale (VAS) in which a respondent selects a whole number (0-10 integers) that best reflects the intensity of his/her pain. Where 0 means no pain and 10 means worst imaginable pain. NPRS was measured at Baseline, 1st Session, 2nd Week and 4th Week
Cranio-vertebral Angle | 40 minutes session, thrice a week for 4 weeks.
  For measuring the angle, the reflective markers will be placed on the tragus of the ear and spinous process of the C7. The camera will be positioned on a tripod 50 cm away from the participant. The axis of the lens of the camera was placed at the level of the shoulder. The photos will be taken and the CVA angle will be calculated by Software Kinovea. CVA was measured at Baseline, 1st Session, 2nd Week and 4th Week
Cervical Joint Position Error Test | 40 minutes session, thrice a week for 4 weeks.
  For measurement of proprioception, Joint Position Error Test is used. The distance/deviation will represent the proprioception deficit (JPE) of each participant. Angle is then calculated by taking arc tan of error distance divided by 90. A meaningful distance of 7.1cm or angle greater than 4.5 degree represents proprioception deficit. JPE Test was measured at Baseline, 1st Session, 2nd Week and 4th Week
Cervical Range of Motion | 40 minutes session, thrice a week for 4 weeks.
  Cervical ROM will be measured by using an inclinometer for Flexion, Extension, Lateral Flexion and Rotation. The normal Range for Flexion is usually approximately 80º. Normal cervical extension is usually 50°, Value for Lateral Flexion is 45° and for rotation its approximately 80°. Cervical ROM were measured at Baseline, 1st Session, 2nd Week and 4th Week

CONTACTS AND LOCATIONS:
Overall Officials: Lal Gul Khan, MScPT, Principal Investigator — Riphah International University
Locations (1):
- Riphah International University, Islamabad, Federal, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dehqan B, Delkhoush CT, Mirmohammadkhani M, Ehsani F. Does forward head posture change subacromial space in active or passive arm elevation? J Man Manip Ther. 2021 Aug;29(4):227-234. doi: 10.1080/10669817.2020.1854010. Epub 2020 Nov 30. PMID 33250012
- [Background] Gonzalez HE, Manns A. Forward head posture: its structural and functional influence on the stomatognathic system, a conceptual study. Cranio. 1996 Jan;14(1):71-80. doi: 10.1080/08869634.1996.11745952. PMID 9086879
- [Background] Kim DH, Kim CJ, Son SM. Neck Pain in Adults with Forward Head Posture: Effects of Craniovertebral Angle and Cervical Range of Motion. Osong Public Health Res Perspect. 2018 Dec;9(6):309-313. doi: 10.24171/j.phrp.2018.9.6.04. PMID 30584494
- [Background] Deshpande V, Bathia K, Kanase S, Pawar A, Jain P, Patel G. Effect of mckenzie approach and neck exercises on forward head posture in young adults. SCOPUS IJPHRD CITATION SCORE. 2019 Jul;10(7):123.
- [Background] Lee MY, Lee HY, Yong MS. Characteristics of cervical position sense in subjects with forward head posture. J Phys Ther Sci. 2014 Nov;26(11):1741-3. doi: 10.1589/jpts.26.1741. Epub 2014 Nov 13. PMID 25435690
- [Background] Ali Ismail AM, Abd El-Azeim AS, El-Sayed Felaya EE. Integrated neuromuscular inhibition technique versus spray and stretch technique in neck pain patients with upper trapezius trigger points: a randomized clinical trial. J Man Manip Ther. 2024 Apr;32(2):141-149. doi: 10.1080/10669817.2023.2192899. Epub 2023 Mar 23. PMID 36951194
- [Background] Khosravi F, Peolsson A, Karimi N, Rahnama L. Scapular Upward Rotator Morphologic Characteristics in Individuals With and Without Forward Head Posture: A Case-Control Study. J Ultrasound Med. 2019 Feb;38(2):337-345. doi: 10.1002/jum.14693. Epub 2018 May 15. PMID 29761537
- [Background] Khan A, Khan Z, Bhati P, Hussain ME. Influence of Forward Head Posture on Cervicocephalic Kinesthesia and Electromyographic Activity of Neck Musculature in Asymptomatic Individuals. J Chiropr Med. 2020 Dec;19(4):230-240. doi: 10.1016/j.jcm.2020.07.002. Epub 2020 Nov 24. PMID 33536860
- [Background] Golzareh S, Shadmehr A, Otadi K, Fereydounnia S. Dry Needling Effects of the Upper Trapezius Muscle on the Angles and Range of Motion of the Neck in Individuals with Forward Head Posture. Journal of Modern Rehabilitation. 2023.
- [Background] Ha SY, Sung YH. A temporary forward head posture decreases function of cervical proprioception. J Exerc Rehabil. 2020 Apr 28;16(2):168-174. doi: 10.12965/jer.2040106.053. eCollection 2020 Apr. PMID 32509702
- [Background] Aggarwal S, Bansal G. Efficacy of integrated neuromuscular inhibition technique in improving cervical function by reducing the trigger points on upper trapezius muscle: A randomized controlled trial. Muller Journal of Medical Sciences and Research. 2018;9(1):1-6.
- [Background] Zalabia M, Abutaleb EE, Diab R, editors. Addition of integrated neuromuscular inhibition technique to amultimodal treatment program for chronic non specific neck pain. International Scientific Conference Faculty of Physical Therapy; 2018.